CLINICAL TRIAL: NCT05844436
Title: Expanded Access Intermediate Size Treatment Protocol: Pritelivir for Immunocompromised Subjects with Treatment Resistant Herpes Simplex Virus Type 1 or 2
Status: Available | Type: Expanded Access
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Collaborators: Impatients N.V. trading as myTomorrows (Industry)
Responsible Party: Sponsor
Other Study IDs: AIC316-03-E-01
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: HSV
MeSH Terms: interventions — pritelivir

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Pritelivir — Participants receive a loading dose of 400 mg (4 x 100 mg tablet) pritelivir on first day followed by continuous dose of 100 mg per day.

SUMMARY:
AiCuris Anti-infective Cures AG (AiCuris) is developing pritelivir for the oral treatment of acyclovir-resistant (ACV-R) mucocutaneous herpes simplex virus (HSV) infections in immunocompromised subjects.

The purpose of the expanded access program (EAP) is to provide pritelivir to immunocompromised subjects with treatment resistant HSV type 1 or 2 who cannot participate in a clinical trial and for whom no approved treatment option is available.

In view of the available pre-clinical and clinical data for pritelivir in immunocompromised subjects with treatment resistant HSV, the lack of treatment options, and the demand for compassionate use of pritelivir, AiCuris aims to provide access to pritelivir via this expanded access program (intermediate size treatment protocol) in the USA. The patient population is focused on those immunocompromised subjects that are not responding to the available FDA-approved antiviral options or cannot use these because of an underlying medical condition. This EAP enables pritelivir to be available as a treatment option for immunocompromised subjects with treatment-resistant HSV type 1 or 2, who do not have access to clinical trial options.

DETAILED DESCRIPTION:
This is a multicenter EAP (via intermediate size treatment protocol) designed to provide access to pritelivir for eligible immunocompromised subjects that are not responding to the available FDA-approved antiviral options or cannot use these because of an underlying medical condition, and who cannot enter a clinical trial. The program will continue until pritelivir becomes available through other mechanisms, or until Sponsor chooses to discontinue the program.

Each subject considered for the EAP will undergo minimal assessment at baseline for lesion assessment and safety (laboratory tests and general physical evaluation). After eligibility check and starting the treatment, the subjects will be monitored on a weekly basis.

ELIGIBILITY:
Main Inclusion Criteria:

1. Immunocompromised (due to conditions including but not limited to HIV infection, hematopoietic-cell or solid organ transplantation, and chronic use of immunosupressive treatment) men and women of any ethnic group aged ≥16 years.
2. ACV-resistant and foscarnet-resistant/intolerant mucocutaneous HSV infection based on clinical failure (no improvement after oral or iv doses for at least 7 days at doses equivalent to or greater than the local agency approved high doses of valacyclovir or famciclovir and/or foscarnet iv therapy or intolerance to foscarnet requiring cessation of foscarnet treatment) or result from genotypic/phenotypic testing or ACV-resistant and previously treated in PRIOH-1 Part C.
3. The current lesion(s) should be confirmed to be positive for HSV before the start of treatment. If not tested beforehand, a lesion swab should be taken for PCR or cell culture before starting treatment, but treatment may be started before obtaining results.
4. Visual confirmation of lesion at start of treatment (including by endoscopy).
5. Willing to remain abstinent or use highly effective method of contraception.
6. Negative pregnancy test for females of childbearing potential at Day 1 and every 4 weeks thereafter.
7. Patient must be willing and able (in the opinion of the physician) to understand the informed consent form.
8. Patient must give written informed consent.

Main Exclusion Criteria:

1. Eligibility and feasibility for a patient to participate in a currently ongoing clinical trial with pritelivir.
2. Known intolerance to pritelivir or any of the excipients (microcrystalline cellulose, croscarmellose sodium, mannitol, colloidal anhydrous silica, magnesium stearate, hydroxy propyl methyl cellulose, polyethylene glycol, calcium diphosphate).
3. Need to use the following medications at any dose: esomeprazole, rabeprazole. Need to use the medications with the following daily dose levels: omeprazole > 20 mg/d, lansoprazole > 20 mg/d or pantoprazole > 80 mg/d.
4. Baseline safety laboratory abnormalities:

   1. ANC < 1000 cells/mm3
   2. Platelet count < 25,000 cells/mm3
   3. Hemoglobin < 8.0 g/dL
   4. AST or ALT > 5 x ULN
   5. Bilirubin > 2.5 x ULN
5. History or current evidence of gastrointestinal malabsorption which, in the opinion of the physician, may affect the extent of absorption of pritelivir.
6. Hemodialysis for any indication and ESRD (eGFR <15 mL/min; stage 5 CKD).
7. History or current evidence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrinological, metabolic, neurological, psychiatric, or other diseases, which, in the opinion of the physician, may affect the patient's safety.
8. Abnormalities in hematological, clinical chemical or any other laboratory variables regarded as clinically relevant by the physician unless they are due to underlying disease or condition.
9. Not able to communicate meaningfully with the physician and site staff.
10. Any other condition which in the opinion of the physician would interfere with successful completion of the treatment.
11. Pregnant and/or breastfeeding women.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult